CLINICAL TRIAL: NCT05442216
Title: Phase II Study of TAGraxofusp and Azacitidine With Venetoclax in Newly Diagnosed Secondary AML After Previous Exposure to HypOmethylatiNG Agents
Brief Title: Tagraxofusp and Azacitidine With Venetoclax in Newly Diagnosed Secondary AML After Hypomethylating Agents
Acronym: TAGALONG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua Zeidner (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Joshua Zeidner, Sponsor Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN AML20-472
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tagraxofusp; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Each treatment cycle will last 28 days. For Cycle 1, tagraxofusp 9 mcg/kg IV over 15 minutes daily for 3 consecutive days followed by azacitidine administered at 75 mg/m2 SQ or IV daily on Day 4 through Day 10. Venetoclax with ramp-up dosing on Day 4 through Day 24. A bone marrow biopsy (BM Bx) will be performed on Day 24 (+3 days) of Cycle 1. If a CRm is obtained, the subject will move to the Continuation Phase. Subjects who do not achieve a CRm will proceed with the next cycle of Induction Phase study treatment.
  Cycle 2+ will consist of tagraxofusp 9 mcg/kg IV over 15 minutes daily (Day 1-3), azacitidine 75 mg/m2 SQ or IV on Day 1 through Day 7 or Days 1-7 or 1-5, 8-9 and venetoclax 400 mg daily Day 1 through Day 21. BM Bx will be performed on Day 21 (+3 days) of Cycle 2. If a CRm is obtained or maintained, the subject will move to or remain on the Continuation Phase. If a CRm is not obtained after Cycle 4, study treatment will be discontinued and the subject will move to follow up
  Interventions: Drug: Tagraxofusp; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Tagraxofusp — 9 mcg/kg intravenously Days 1-3
Drug: Azacitidine — 75 mg/m2 subcutaneously or intravenously Days 1-7
Drug: Venetoclax — 400 mg daily Days 1-21.

SUMMARY:
A treatment cycle is 28 days. Tagraxofusp will be administered at 9 mcg/kg IV over 15 minutes (-5 or +15 minutes) daily for 3 consecutive days (or 3 doses over a period not to exceed 10 days if postponement is required to allow for toxicity resolution), followed by azacitidine administered at 75 mg/m2 SQ or IV daily on Day 4 through Day 10. Venetoclax will begin on Day 4 and continue through Day 24 (21 consecutive days). A bone marrow biopsy (BM Bx) will be performed on Day 24 (+3 days) of Cycle 1.

Subjects who do not achieve a CRm will proceed with the next cycle of Induction Phase study treatment, irrespective of hematologic laboratory values. Cycle 2+ will consist of tagraxofusp 9 mcg/kg IV over 15 minutes daily for 3 consecutive days (Day 1-3 or 3 doses over a period not to exceed 10 days if postponement is required to allow for toxicity resolution), azacitidine 75 mg/m2 SQ or IV on Day 1 through Day 7 or Days 1-7 or 1-5, 8-9 and venetoclax 400 mg daily Day 1 through Day 21.

A bone marrow biopsy (BM Bx) will be performed on Day 21 (+3 days) of Cycle 2. If a CRm is obtained or maintained, the subject will move to or remain on the Continuation Phase. Subjects who do not achieve a marrow CR (CRm) after Cycle 2 will proceed with the next cycle of Induction Phase study treatment as described above, irrespective of hematologic laboratory values. If a CRm is obtained after Cycle 3 or 4, the subject will move to the Continuation Phase .

If a CRm is not obtained after Cycle 4, study treatment will be discontinued and the subject will move to follow up. If per the investigator, the subject is receiving clinical benefit, study treatment may continue until toxicity or completion of 12 total cycles. A BM Bx will be performed at least every 3 cycles for these subjects.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Subjects must have newly diagnosed, untreated AML, as defined by ≥ 20% blasts in peripheral blood or bone marrow by manual aspirate differential, immunohistochemistry staining, or flow cytometry, as defined by standard WHO 2016 diagnostic criteria.
* Subjects must have documented CD123 positivity on leukemia cells by a centralized flow cytometry assay (Hematologics).
* Documented diagnosis of prior MDS, CMML, MDS/MPN overlap syndromes, or MPN's according to WHO criteria. Subjects must have received at least 2 cycles of hypomethylating agents (azacitidine or decitabine or oral decitabine/cedazuridine) for the management of MDS, CMML, MDS/MPN overlap syndromes, or MPN's. NOTE: Subjects who have enrolled on clinical trials with investigational agents in combination with HMA's will still be eligible. Investigational agents must have been discontinued >14 days prior to study treatment initiation. Subjects who have enrolled on clinical trials with investigational agents in combination with HMA's will still be eligible. Investigational agents must have been discontinued > 21 days prior to study treatment initiation.
* WBC < 30 x 109 /µL- subjects with WBC ≥ 30 x 109 /µL may still be eligible after receiving cytoreduction measures such as hydroxyurea, and/or leukapheresis, if WBC < 30 x 109 /µL prior to study treatment initiation. Cytoreduction with hydroxyurea, leukapheresis and/or cyclophosphamide is allowed prior to treatment. Hydroxyurea must be discontinued ≥ 12 hours prior to study treatment initiation. Cyclophosphamide must be discontinued ≥ 5 days prior to study treatment initiation.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-2.
* Demonstrate adequate organ function within 28 days prior to registration.
* Left ventricular ejection fraction (LVEF) ≥ 45%.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential and male participants must be willing to use effective contraception as outlined in the protocol.
* Known HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* Patients with known evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Subjects who are suitable for and are willing to receive intensive chemotherapy.
* Diagnosis of acute promyelocytic leukemia.
* Known CNS involvement with AML.
* Previous receipt of tagraxofusp.
* Treatment with chemotherapy, wide-field radiation, or biologic therapy within 14 days of registration. NOTE: hydroxyurea, leukapheresis and/or cyclophosphamide are allowed prior to study entry per the protocol.
* Treatment with investigational drug within 21 days of registration.
* Previous allogeneic stem cell transplant within 60 days prior to registration.
* Receiving immunosuppression therapy, with the exception of prednisone ≤ 10mg/d, for the treatment or prophylaxis of GVHD. If the patient has been on immunosuppressant treatment or prophylaxis for GVHD, the treatment must have been discontinued at least 14 days prior to study treatment initiation and there must be no evidence of Grade ≥ 2 GVHD.
* History of other malignancies (excluding MDS, CMML, MDS/MPN, MPN's) within 2 years prior to reigstration, with the exception of: adequately treated in situ carcinoma of the cervix, breast, prostate; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent. Subjects receiving maintenance or adjuvant therapy for organ-confined malignancy such as breast or prostate cancer are eligible. Maintenance and/or adjuvant chemotherapy must be discontinued >72 hours prior to study treatment initiation. Those with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the sponsor-investigator before registration.
* Clinically significant cardiovascular disease including:

  * Uncontrolled CHF
  * Cardiac insufficiency Grade III or IV per New York Heart Association (NYHA) classification
  * Uncontrolled angina/hypertension/arrhythmia
  * Clinically significant abnormalities on a 12-lead electrocardiogram
  * History of myocardial infarction or stroke within 6 months of registration
* Uncontrolled significant pulmonary disease (e.g., COPD, pulmonary hypertension) that in the opinion of the investigator would put the patient at significant risk for pulmonary complications during the study.
* Active uncontrolled or severe systemic infection. Enrollment is possible after control of infection, at discretion of the treating physician.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Other severe medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, and in the judgement of the investigator would make the patient inappropriate for enrollment in this study. This may include psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 5 years
  The CR rate based on ELN AML response criteria in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax

SECONDARY OUTCOMES:
Assess adverse events | 4 months
  Describe overall toxicity of tagraxofusp and azacitidine and venetoclax. The frequency and nature of adverse events will be assessed by NCI CTCAE v5.0.
Rate of CR + CRh | 5 years
  Estimate the rate of CR + CRh in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax.The rate of CR + CRh is defined as bone marrow myeloblasts of < 5% combined with both absolute neutrophil count > 500/μL and platelet count > 50 × 109/L.
Rate of CR without evidence of Minimal Residual Disease (MRD) | 5 years
  CR without evidence of MRD in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax based on ELN AML response criteria.
Overall Response Rate (ORR) | 5 years
  Estimate the ORR in patients with newly diagnosed AML with p-HMA who receive tagraxofusp and azacitidine and venetoclax. ORR (partial remission [PR] + CR + CRi + morphological leukemia-free state [MLFS]) as defined by ELN-2017.
Overall Survival (OS) | 5 years
  Estimate OS in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax. OS is defined as time from initiation of treatment until death or last follow-up.
Disease Free Survival (DFS) | 5 years
  Estimate the DFS in subjects with newly diagnosed AML with p-HMA after receiving tagraxofusp and azacitidine and venetoclax. DFS is defined as time from CR/CRi until relapse, death, or last follow-up, as based on ELN-2017.
Recurrence Free Survival (RFS) | 5 years
  Estimate the recurrence free survival (RFS) in subjects with newly diagnosed AML with p-HMA after receiving tagraxofusp and azacitidine and venetoclax. RFS is defined as time from ORR until progression, relapse, or death. Subjects who have not progressed will be right-censored at the date of the last disease evaluation.
Event-Free Survival (EFS) | 5 years
  Estimate the event-free survival (EFS) in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax. EFS is defined as time from initiation of treatment until no response (after 2 cycles of tagraxofusp), relapse or death.
Rate of allogeneic stem cell transplant | 4 months
  Estimate the rate of allogeneic stem cell transplant in subjects with newly diagnosed AML with p-HMA receiving tagraxofusp and azacitidine and venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Zeidner, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (7):
- United States (7):
  - University of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Penn Medicine Abramson Cancer Center, Philadelphia, Pennsylvania
  - Lifespan Health System Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No